CLINICAL TRIAL: NCT02790398
Title: Transdiagnostic Up-regulation of Positive Affect in Emotional Disorders: A Randomized Pilot Study
Brief Title: Up-regulating Positive Affect in Emotional Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaumeI_Transd_PS
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-03

CONDITIONS: Anxiety; Depression
Keywords: Transdiagnostic treatment protocol; Transdiagnostic treatment protocol + PA component
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdiagnostic treatment protocol (Experimental): Transdiagnostic treatment protocol.
  Interventions: Behavioral: Transdiagnostic treatment protocol
- Transdiagnostic treatment protocol + PA regulation component (Active Comparator): Transdiagnostic treatment protocol that includes a component aimed at the regulation of PA.
  Interventions: Behavioral: Transdiagnostic treatment protocol + PA regulation component

INTERVENTIONS:
Behavioral: Transdiagnostic treatment protocol — Transdiagnostic treatment protocol for emotional disorders whose aims are to learn and practice adaptive ways to regulate emotions from a transdiagnostic perspective. The protocol contains the following components: present-focused emotional awareness, cognitive flexibility, emotional avoidance and emotion driven behaviors, interoceptive and situation-based emotion exposure, psychoeducation about emotions, motivational enhancement and relapse prevention. These components are organized in twelve modules.
  Arms: Transdiagnostic treatment protocol
Behavioral: Transdiagnostic treatment protocol + PA regulation component — Transdiagnostic treatment protocol for emotional disorders + PA regulation components has the purpose of learning and practicing adaptive ways to regulate emotions from a transdiagnostic perspective. This protocol includes the same components but it also includes 4 additional modules focused specifically on the regulation of positive affectivity.
  Arms: Transdiagnostic treatment protocol + PA regulation component

SUMMARY:
The aim of this study is to assess the differential effect of two transdiagnostic treatment protocols for emotional disorders (ED) (depression and anxiety disorders) using a randomized pilot study design: a) a transdiagnostic treatment protocol (TTP) based on the Unified Protocol; and b) a version of this protocol that also includes a specific component to address the regulation of positive affect (TTP+PA). Another aim was to assess the acceptability of both treatments by patients. It was hypothesized that the intervention would result in significant differences in favor of the TTP+PA protocol in all measures. Regarding acceptability, it was hypothesized that both treatments (TP and TP+PA) would be well-accepted by the two groups of participants.

DETAILED DESCRIPTION:
ED are highly prevalent mental disorders and one of the main causes of disability worldwide. Currently, there is evidence showing the efficacy of transdiagnostic treatments for anxiety disorders, and for comorbid depression and anxiety disorders. An important line of research within the transdiagnostic treatment of ED was initiated by D. H. Barlow. Barlow's theory of triple vulnerability emphasizes the underlying vulnerabilities that are common to ED and help to explain the comorbidity among these diverse conditions. A central aspect within this theoretical perspective is the role of emotion regulation in ED. The regulation of negative emotions in ED has received a great deal of attention in cognitive behavior therapy (CBT) research, and more recently in transdiagnostic ED models like the UP developed by Barlow's team. However, although Barlow underscored the role of low PA in the onset and maintenance of ED, the main objective of the treatment components in the UP is to train patients in negative affect (NA) regulation, but less attention has been paid to the inclusion of treatment components to directly target PA regulation. Moreover, literature has shown that higher levels of PA are associated with better physical and psychological health, healthier lifestyles, and better general functioning. Consequently, an important treatment goal from a transdiagnostic treatment approach would be to increase PA while decreasing NA.

The aim of this study is to compare the differential effect of two transdiagnostic treatment protocols for ED using a randomized pilot study design: a) a transdiagnostic treatment protocol (TTP) based on the Unified Protocol; and b) a version of this protocol that also includes a specific component to address the regulation of positive affect (TTP+PA). Another aim is to assess the acceptability of both treatments by patients. It was hypothesized that the intervention would result in significant differences in favor of the TTP+PA protocol in all measures. Regarding acceptability, it was hypothesized that both treatments (TP and TP+PA) would be well-accepted by the two groups of participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* meeting the DSM-IV diagnostic criteria for ED (major depression disorder, dysthimic disorder, generalized anxiety disorder, social anxiety disorder, panic disorder, agoraphobia, obsessive-compulsive disorder, anxiety disorder not otherwise specified, unipolar mood disorder not otherwise specified)
* ability to understand and read Spanish

Exclusion Criteria:+

* bipolar disorder
* schizophrenia
* risk of suicide
* receiving another psychological treatment during the study
* in the case of receiving pharmacological treatment, an increase and/or change in this treatment during the study period (a decrease in pharmacological treatment is accepted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in the Positive and Negative Affect Scale (PANAS) at pre-, post-intervention (up to 4 months) and at 3-month follow-up. | Up to 7 months
  The PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is from 10 to 50. The Spanish version has demonstrated high internal consistency (α = 0.89 and 0.91 for PA and NA in women, respectively, and α = 0.87 and 0.89 for PA and NA in men, respectively) in college students.

SECONDARY OUTCOMES:
Change in the Beck Depression Inventory II (BDI-II) at pre-, post-intervention (up to 4 months) and at 3-month follow-up. | Up to 7 months
  The BDI-II is one of the most widely used questionnaires to evaluate the severity of depression in pharmacological and psychotherapy trials. It consists of 21 items about the different symptoms characterizing the major depression disorder, summed to obtain the total score, which can be a maximum of 63 points. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and a test-retest reliability of around 0.8.
Change in the Overall Anxiety Severity and Impairment Scale (OASIS) at pre-, post-intervention (up to 4 months) and at 3-month follow-up. | Up to 7 months
  The OASIS consists of a 5-item questionnaire, rated from 0 to 4, that assesses the frequency and severity of the anxiety symptoms. The instrument also provides measures of avoidance, as well as work, academic, social and everyday life impairment related to anxiety symptoms. A psychometric analysis of the OASIS scale found good internal consistency (α = .80), test-retest reliability (k = .82) and convergent validity for this instrument.
Change in the Quality of Life Inventory (QLI) at pre-, post-intervention (up to 4 months) and at 3-month follow-up. | Up to 7 months
  The QLI is a brief self-report questionnaire that assesses perceived quality of life in different life-related areas. The questionnaire includes 10 items, rated on a scale from one to 10, that assess physical well-being, psychological well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, social emotional support, community and services support, personal fulfillment, spiritual fulfillment and overall quality of life. The QLI has shown excellent internal consistency (between .90 and .92), test-retest reliability (.87) and discriminant validity. The Spanish validation of the QLI has also demonstrated good test-retest reliability (α = .89) and discriminant validity.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Gonzalez-Robles, PhD student, Study Chair — Universitat Juame I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No